CLINICAL TRIAL: NCT04223869
Title: Critical Role of Interleukin-34 in Gingival Crevicular Fluid as a Potential Markers of Inflammation in Patients With Periodontitis
Brief Title: IL-34 Levels in Various Types of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Seyma Bozkurt Doğan, Associate Professor, Ankara Yildirim Beyazıt University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-106-03/06
Record Dates: First submitted 2020-01-08; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Chronic Periodontitis; Aggressive Periodontitis
Keywords: Periodontitis; Interleukin 34; RANKL; OPG; gingival crevicular fluid
MeSH Terms: conditions — Chronic Periodontitis; Aggressive Periodontitis; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- periodontally healthy group (No Intervention): Control
- Chronic Periodontitis (Active Comparator): non-surgical periodontal treatment was performed
  Interventions: Other: non-surgical periodontal treatment
- Aggressive Periodontitis (Active Comparator): non-surgical periodontal treatment was performed
  Interventions: Other: non-surgical periodontal treatment

INTERVENTIONS:
Other: non-surgical periodontal treatment — scaling and root planing were performed
  Arms: Aggressive Periodontitis; Chronic Periodontitis

SUMMARY:
The objective of this study is to 1) identification of the impact of IL-34 on the pathogenesis of periodontal disease and determine whether any relationship among the existing levels of Gingival crevicular fluid (GCF) Interleukin 34( IL-34 )and GCF Receptor activator of nuclear factor -kB ligand (RANKL), osteoprotegerin (OPG) and RANKL/OPG ratio, as a mediator of bone resorption 2) analysis of the impact of non-surgical periodontal treatment on GCF IL-34 levels in patients with chronic periodontitis (CP) and aggressive periodontitis (AgP) and 3) to correlate between biochemical markers and clinical recordings

DETAILED DESCRIPTION:
A novel cytokine interleukin 34 (IL-34) is a second possible functional ligand of macrophage colony-stimulating factor-1 receptor (CSF-1R). IL-34 is secreted in different tissues including: heart, brain, lung, liver, kidney, thymus, testes, ovary, small intestine, prostate, colon and spleen . IL-34 shares vital functions of macrophage colony-stimulating factor -1(CSF-1), and manage myeloid cell survival, differentiation and proliferation. It is produced by synovial fluid, gingival fibroblast and human adipose tissue, and is controlled by the transcription factor RANK and activation of c-Jun N-terminal kinase (CJNK). Additionally, the pro-inflammatory cytokines tumornecrosis factor-alfa (TNF-α) and interleukin-1beta (IL-1β) arrange IL-34 release from gingival fibroblasts, by a mechanism including nuclear factor -kB (NF-kB) and mitogen activated protein kinase (MAPK).The targeting CSF-1 merely is not adequate to inhibit the effect via CSF-1R. Moreover, neither RANKL nor IL-34 solely can cause osteoclast formation which suggests that IL-34 is required but not enough. IL-34 plays a crucial role in RANKL-induced osteoclastogenesis; the osteoclasts differentiation is mediated by the same way with CSF-1.

Several studies evaluated the role of IL-34 in the pathogenesis of chronic periodontitis (CP). To the best of our knowledge, any of these studies reported the relationship between GCF IL-34 level and GCF RANKL/OPG ratio in other types of periodontitis before and after non-surgical periodontal therapy. This study highlights the influence of IL-34 in the pathogenesis of Chronic Periodontitis (CP) and Aggressive Periodontitis (AgP).

The objective of this study is to 1) identification of the impact of IL-34 on the pathogenesis of periodontal disease and determine whether any relationship among the existing levels of GCF IL-34 and GCF RANKL, OPG and RANKL/OPG ratio, as a mediator of bone resorption 2) analysis of the impact of non-surgical periodontal treatment on GCF IL-34 levels in patients with CP and AgP and 3) to correlate between biochemical markers and clinical recordings.

The study included 60 subjects: 20 who were periodontally healthy (CTRL), 20 with chronic periodontitis (CP)and 20 with aggressive periodontitis (AgP). Patients with periodontitis were treated with non-surgical periodontal therapy. GCF sampling procedures and clinical periodontal measures were investigated at the baseline and 6 weeks after treatment. Levels of IL-34, RANKL and OPG were analyzed with Enzyme-linked immunosorbent assay (ELISA).

Participants were periodontally assessed at baseline and after non-surgical periodontal therapy in accordance with the following criteria; plaque index (PI)(Silness and Loe, 1964), GI(Loe and Silness, 1963), PPD, clinical attachment level (CAL) and BOP (judged positive if it developed within 15 s following contact). Full-mouth periapical radiographs were used to determine the periodontal bone loss.The clinical measurement were taken in millimeters by a single calibrated examiner (ŞBD), who was blinded to the whole study composition, from six locations of each tooth (mesio-buccal, disto-buccal, mid-buccal, mesiolingual, disto-lingual, and mid-lingual), by the use of a periodontal probe (Hu-Friedy, Chicago, IL, USA).

Two sites per participant were selected to collect GCF for each group. GCF samples were collected from the mesiobuccal or distobuccal sites of single-rooted teeth. The sample areas were isolated with cotton rolls, saliva contamination was ensured, all supragingival plaque was eliminated by sterile curette and it was slightly air dried. The paper strips were inserted within the crevice until resistance was encountered and then allowed to remain in place for 30 seconds. The amount of GCF on the strips was measured by weighing the collected liquid. The strips were placed into closed and numbered plastic eppendorf tubes. The liquid was weighed again, immediately after collection, to take into account evaporation. The samples consisting of saliva and blood were discarded from the study. Two available for use samples from per individual were merged to make a singular sample and instantly insert in a singular Eppendorf tube and freezed at _80°C until aftertime evaluation.

ELIGIBILITY:
Inclusion Criteria:

* CP group included 20 patients, ≥ 35 years of age, and this category was displayed as a minimum of six teeth available clinical attachment loss (AL) and pocket probing depth (PPD) ≥ 5mm. These teeth exhibited positive bleeding on probing (BOP) across a minumum 2 separate quadrants and bone loss affecting >30 % of available teeth on clinical and radiographic inspection. The gingival index (GI) score for indications of inflammation (red color and edema of the gingival margin) was >1 for the CP group.
* AgP group included 20 patients, <35 years of age, and cases showed PPD≥ 5mm with at least six teeth and radiographic evidence of alveolar bone loss. At least three of these six teeth with PPD ≥ 5 mm were not molars or incisors. These patients showed severe periodontal tissue devastation and decrease of periodontal support conflicting with age and plaque levels.
* Control group included 20 participants and they presented PPD ≤ 3mm, GI=0 (nonavailable of clinical inflammation), absence of alveolar bone loss (e.g., distance between the cemento-enamel junction and the bone crest was <3mm in> 95% of proximal tooth sites).
* All participants had minimum 20 teeth and their overall systematic health

Exclusion Criteria:

* lactation
* pregnancy
* current and ex-smoking habits
* undergone nonsurgical periodontal therapy and prescription of antibiotics or non-steroidal anti-inflammatory medication within the previous 6 months or surgical periodontal treatment within the preceding year
* postmenopause
* systemic conditions such as; diabetes mellitus, cancer, cardiovascular and respiratory diseases, rheumatoid arthritis, osteoporosis, or immunologic disorders, that might cause progress of periodontal disease.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
gingival crevicular fluid IL-34 level | 6th week
  gingival crevicular fluid IL-34 levels change from baseline to at 6th week

SECONDARY OUTCOMES:
Gingival crevicular fluid RANKL level | 6th week
  change of gingival crevicular fluid RANKL levels from baseline at 6th weeks
Gingival crevicular fluid OPG level | 6th week
  change of gingival crevicular fluid OPG levels from baseline at 6th weeks
Plaque index | 6th week
  oral hygiene score
Gingival index | 6th week
  gingival inflammation score
bleeding on probing | 6th week
  deemed positive if it occurred within 15 seconds after probing
clinical attachment level | 6th week
  distance between the cemento-enamel junction to the deepest point of periodontal pocket

CONTACTS AND LOCATIONS:
Overall Officials: Umut Ballı, PhD, DDS, Principal Investigator — Bülent Ecevit University Faculty of Dentistry; Figen Öngöz Dede, PhD, DDS, Principal Investigator — Ordu University; Şeyma Bozkurt Doğan, PhD, DDS, Study Chair — Ankara Yildirim Beyazıt University; Erdim Sertoğlu, PhD, DDS, Principal Investigator — Ankara Sağlık Bilimleri University